CLINICAL TRIAL: NCT04707716
Title: Implant Supported Single Crowns With Different Retention Modes - Effects on Peri-implant Tissue: A Prospective Randomized Controlled Clinical Trial
Brief Title: Implant Supported Single Crowns With Different Retention Modes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32-578 ex 19/20
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Complications: Inflammatory Reactions, Mechanical Complications
Keywords: MMP-8; marginal bone level; conometric concept - Acuris; crown retention; all-ceramic crown
MeSH Terms: interventions — Cementation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conometric concept (Acuris system) (Experimental): single implant crown retention using friction only
  Interventions: Other: conometric concept Acuris system
- screw retention (Active Comparator): screw retained implant Crown fixation
  Interventions: Other: screw retention
- cementation (Active Comparator): cement retained implant Crown fixation
  Interventions: Other: cementation

INTERVENTIONS:
Other: conometric concept Acuris system — implant crown retention type using friction only
  Arms: conometric concept (Acuris system)
Other: screw retention — screw retained implant crown
  Arms: screw retention
Other: cementation — cement retained implant crown
  Arms: cementation

SUMMARY:
This study aims to examine the inflammatory response mediated by MMP-8 (Matrix metalloproteinase-8 ) level in peri-implant sulcus fluid adjacent to screw-retained, cemented or using the Acuris-system fixed single implant crowns as well as changing of the marginal bone level within the first year after implant restoration. Furthermore periodontal parameters, patient satisfaction and possible occurring biological or technical complications will be evaluated.

DETAILED DESCRIPTION:
After giving their written consent volunteers will be screened and eligible subjects will be randomized to three different groups. In group 1 Acuris® is used as fixation type; in group 2 screw retention, and in group 3 cementation is used. After 3 months of submerged healing the dental implants will be restored with all ceramic single implant crowns, fixed by using the randomized fixation mode. Follow-up visits till one year after implant restoration will be performed. At least 11 study visits during 16 months will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* capability of giving an informed consent
* good health as defined by the subjects medical history (no contraindications as described in the exclusion criteria below)
* age 18 to 99 years
* Good periodontal status: BOP < 20%, PI < 30%, no PD > 4mm
* No heavy smokers (< 10 cigarettes/day)
* at least 1 missing tooth in the premolar and molar region (with at least a mesial neighboring tooth/implant showing adequate hard- and soft tissue situation without the need of crestal hard- or soft tissue augmentation) either in the maxilla or in the mandible requiring implant therapy for reconstruction, requiring sinus floor augmentation or not.

Exclusion Criteria

* Insufficient bone volume for implant placement requiring GBR (guided bone regeneration) procedure in crestal area.
* Heavy Smokers (>10 cigarettes/day)
* Medication with a contraindication for implant therapy (especially antiresorptive therapy, ongoing or recently completed local radiotherapy, systematic diseases, ongoing immunosuppressive therapy, functional disorders like Bruxism).
* Skeletal immaturity.
* Any active malignancy or ongoing treatment for malignancy.
* An active infection (e.g. caries, gingivitis, periodontitis) at or in the neighboring area of the operative site.
* Pregnancy
* unable or unwilling to return for follow-up visits for a period of at least 16 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Change of marginal bone level | at baseline, 4 months after implant placement and 3, 6 and 12 months after restoration
  assessed by single tooth x-ray; in mm
Change of matrix metalloproteinase 8 level | 4 months after implant placement, 3, 6 and 12 months after integration of the implant crown
  biomarker for Inflammation of peri-implant disease; in ng/ml

SECONDARY OUTCOMES:
Change of probing depth (PD) | at baseline, 4, 7, 10, 16 months after implantation
  using a periodontal probe; in mm
Number of occurrences of chipping | measured after integration of implant crown 3, 6 and 12 months after restoration
  visual check
soft tissue maintenance | measured 4 months after implant placement and 3, 6 and 12 months after restoration
  Papilla Index (Jemt T, 1997), the index ranges from 0 to 4, while 2 and 3 indicate physiological outcome
technician satisfaction | measured 12 months after restoration
  evaluated using an individual questionnaire
dentist satisfaction | measured 12 months after restoration
  evaluated using an individual questionnaire
patient satisfaction | measured at baseline, 3 and 12 months after restoration
  evaluated using OHIP-G 14 questionnaire. The following dimensions are captured by the OHIP-G 14: functional Limitation (e.g., "pronouncing any words because of problems with your teeth, mouth, dentures, or jaw?") and physical Pain (e.g., "Have you had painful aching in your mouth"). 14 questions are raised, which are answered using a rating scale from 0 (never) to 4 (very often).
Plaque Index (PI) | at baseline, 4, 7, 10 and 16 months after implantation
  in percent
Bleeding on Probing (BOP) | at baseline, 4, 7, 10 and 16 months after implantation
  in percent
Patient satisfaction concerning the implant crown | measured 12 months after restoration
  evaluated using an individual questionnaire
Number of occurrences of fractures | measured after integration of implant crown 3, 6 and 12 months after restoration
  visual check
Number of occurrences of screw loosening | measured after integration of implant crown 3, 6 and 12 months after restoration
  visual check
Number of occurrences of crown loosening | measured after integration of implant crown 3, 6 and 12 months after restoration
  visual check

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Jakse, UnivProfDDr, Principal Investigator — Department of Dental Medicine and Oral Health
Locations (1):
- Medical University of Graz, Department of Dental Medicine and Oral Health, Division of Oral Surgery and Orthodontics, Graz, Austria

REFERENCES:
- [Background] DeCarlo AA, Grenett HE, Harber GJ, Windsor LJ, Bodden MK, Birkedal-Hansen B, Birkedal-Hansen H. Induction of matrix metalloproteinases and a collagen-degrading phenotype in fibroblasts and epithelial cells by secreted Porphyromonas gingivalis proteinase. J Periodontal Res. 1998 Oct;33(7):408-20. doi: 10.1111/j.1600-0765.1998.tb02337.x. PMID 9842506
- [Background] Jemt T. Regeneration of gingival papillae after single-implant treatment. Int J Periodontics Restorative Dent. 1997 Aug;17(4):326-33. PMID 9497723
- [Background] Kraus RD, Epprecht A, Hammerle CHF, Sailer I, Thoma DS. Cemented vs screw-retained zirconia-based single implant reconstructions: A 3-year prospective randomized controlled clinical trial. Clin Implant Dent Relat Res. 2019 Aug;21(4):578-585. doi: 10.1111/cid.12735. Epub 2019 Mar 12. PMID 30861635
- [Background] Lekholm U, Adell R, Lindhe J, Branemark PI, Eriksson B, Rockler B, Lindvall AM, Yoneyama T. Marginal tissue reactions at osseointegrated titanium fixtures. (II) A cross-sectional retrospective study. Int J Oral Maxillofac Surg. 1986 Feb;15(1):53-61. doi: 10.1016/s0300-9785(86)80011-4. PMID 3083006
- [Background] Lemos CA, de Souza Batista VE, Almeida DA, Santiago Junior JF, Verri FR, Pellizzer EP. Evaluation of cement-retained versus screw-retained implant-supported restorations for marginal bone loss: A systematic review and meta-analysis. J Prosthet Dent. 2016 Apr;115(4):419-27. doi: 10.1016/j.prosdent.2015.08.026. Epub 2015 Nov 14. PMID 26589441
- [Background] Lorenzoni M, Pertl C, Wegscheider W, Keil C, Penkner K, Polansky R, Bratschko RO. Retrospective analysis of Frialit-2 implants in the augmented sinus. Int J Periodontics Restorative Dent. 2000 Jun;20(3):255-67. PMID 11203567
- [Background] Ma J, Kitti U, Teronen O, Sorsa T, Husa V, Laine P, Ronka H, Salo T, Lindqvist C, Konttinen YT. Collagenases in different categories of peri-implant vertical bone loss. J Dent Res. 2000 Nov;79(11):1870-3. doi: 10.1177/00220345000790110901. PMID 11145357
- [Background] Meissen R, Mintcheva M, Netuschil L. Matrix metalloproteinase-8 levels in peri-implant sulcus fluid adjacent to titanium and zirconium nitride surfaces. Int J Periodontics Restorative Dent. 2014 Jan-Feb;34(1):91-5. doi: 10.11607/prd.1504. PMID 24396843
- [Background] Penarrocha-Oltra D, Monreal-Bello A, Penarrocha-Diago M, Alonso-Perez-Barquero J, Botticelli D, Canullo L. Microbial Colonization of the Peri-Implant Sulcus and Implant Connection of Implants Restored With Cemented Versus Screw-Retained Superstructures: A Cross-Sectional Study. J Periodontol. 2016 Sep;87(9):1002-11. doi: 10.1902/jop.2016.160017. Epub 2016 May 6. PMID 27153291
- [Background] Sailer I, Muhlemann S, Zwahlen M, Hammerle CH, Schneider D. Cemented and screw-retained implant reconstructions: a systematic review of the survival and complication rates. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:163-201. doi: 10.1111/j.1600-0501.2012.02538.x. PMID 23062142
- [Background] Sorsa T, Tjaderhane L, Konttinen YT, Lauhio A, Salo T, Lee HM, Golub LM, Brown DL, Mantyla P. Matrix metalloproteinases: contribution to pathogenesis, diagnosis and treatment of periodontal inflammation. Ann Med. 2006;38(5):306-21. doi: 10.1080/07853890600800103. PMID 16938801
- [Background] Sorsa T, Hernandez M, Leppilahti J, Munjal S, Netuschil L, Mantyla P. Detection of gingival crevicular fluid MMP-8 levels with different laboratory and chair-side methods. Oral Dis. 2010 Jan;16(1):39-45. doi: 10.1111/j.1601-0825.2009.01603.x. Epub 2009 Jul 8. PMID 19627514
- [Background] Teughels W, Van Assche N, Sliepen I, Quirynen M. Effect of material characteristics and/or surface topography on biofilm development. Clin Oral Implants Res. 2006 Oct;17 Suppl 2:68-81. doi: 10.1111/j.1600-0501.2006.01353.x. PMID 16968383
- [Background] Thoma DS, Sailer I, Muhlemann S, Gil A, Jung RE, Hammerle CHF. Randomized controlled clinical study of veneered zirconia abutments for single implant crowns: Clinical, histological, and microbiological outcomes. Clin Implant Dent Relat Res. 2018 Dec;20(6):988-996. doi: 10.1111/cid.12674. Epub 2018 Oct 17. PMID 30328283
- [Background] Vindasiute E, Puisys A, Maslova N, Linkeviciene L, Peciuliene V, Linkevicius T. Clinical Factors Influencing Removal of the Cement Excess in Implant-Supported Restorations. Clin Implant Dent Relat Res. 2015 Aug;17(4):771-8. doi: 10.1111/cid.12170. Epub 2013 Nov 14. PMID 24224895